CLINICAL TRIAL: NCT06776393
Title: Longitudinal Non-invasive Analysis of VOCAle Cord Function Based on Trans-laryngeal Ultrasound Acquisitions and Voice Recordings
Acronym: VOCALISE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP240029
Record Dates: First submitted 2024-10-23; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-10

CONDITIONS: Postoperative Dysphonia
Keywords: motion mode ultrasound; voice recordings; GRBASI scale; VHI
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Intervention Model Description: patients who have undergone cervical endocrine surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients diagnosed with dysphonia following cervical endocrine surgery (Other): Prospective single-center cohort study in patients diagnosed with dysphonia following cervical endocrine surgery
  Interventions: Other: ultrasound

INTERVENTIONS:
Other: ultrasound — "Dynamic translaryngeal Ultrasound Motion mode ultrasound of the laryngeal region during phonation Acoustic recordings VHI questionnaires "
  Other Names: voice recordings

SUMMARY:
The main objective of VOCALISE study is to propose a new approach allowing a better characterization of postoperative dysphonia. This involves associating with dynamic translaryngeal ultrasound optimized acquisitions of the vibration of each vocal fold in phonation simultaneously with voice recordings. A software program to analyze the displacement of arytenoids, markers of substitution of the vocal cords, will be developed to finely quantify the mobility of laryngeal structures, by combining classical methods of motion analysis and deep learning methods.

This approach will be evaluated to follow speech therapy rehabilitation in patients with post-operative dysphonia following recurrent nerve injury.

DETAILED DESCRIPTION:
Dynamic translaryngeal ultrasound (dTLUS), a non-invasive and inexpensive technique, has emerged in recent years as an alternative to nasofibroscopy for assessing vocal cord paralysis. This paralysis is the major risk (3 to 5%) associated with cervical surgery (100,000 procedures per year in France). Initial work by our consortium has demonstrated the performance of dTLUS after thyroid or parathyroid surgery in the early diagnosis of vocal cord paralysis. The aim of VOCALISE is to propose a new approach for better characterisation of post-operative dysphonia. This involves combining optimised dTLUS acquisitions with acquisitions of the vibration of each vocal cord during phonation, simultaneously with voice recordings. Software will be developed to analyse the displacement of the arytenoids, which are surrogate markers for the vocal cords, in order to quantify the mobility of laryngeal structures in fine detail, using a combination of conventional motion analysis methods and deep learning methods.

This approach will be evaluated to monitor speech therapy rehabilitation in patients with post-operative dysphonia following a lesion of the recurrent nerve.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* Obtaining patient's free and informed consent
* Patients with dysphonia following cervical surgery and referred for speech therapy
* Social security scheme membership (beneficiary or entitled), excluding MA

Exclusion Criteria:

* Known preoperative history of recurrent nerve paralysis (PR)
* History of laryngeal or vocal cord tumour
* Surgical complications preventing proper assessment of postoperative vocal cord mobility (tracheotomy, tracheal resection).
* Patients with a history of thyroid or parathyroid surgery or cervicotomy for another pathology
* Patient under guardianship or guardianship or deprived of liberty or under safeguard of justice
* Pregnant or nursing patient
* Patient does not read or has vision problems
* Cognitive and/or auditory impairment preventing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the contribution of translaryngeal ultrasound combined with acoustic and perceptual measurements of voice and speech classically used in speech therapy for the rehabilitation of patients with dysphonia following surgery. | 6 months
  Correlation of each quantitative evaluation criterion proposed in ultrasound and voice and speech analysis with the classical voice quality criteria: the VHI (voice handicap index), the GRBASI scale (defined by 5 expert speech pathologists) and a set of acoustic measures of voice and speech.

SECONDARY OUTCOMES:
To visualise arytenoid motion in subjects with shadow artifact using the standard dTLUS approach, by optimising dTLUS acquisitions including curvilinear probe acquisitions, gel cushion acquisitions and lateral mode acquisitions. | 6 months
  - Correlation between spectral measurements made with ultrasound in motion mode with spectral measurements obtained from voice recording.
To visualise arytenoid motion in subjects with shadow artifact using the standard dTLUS approach, by optimising dTLUS acquisitions including curvilinear probe acquisitions, gel cushion acquisitions and lateral mode acquisitions. | 6 months
  - Comparison of spectral measurements made in M mode on the left and right sides in two groups of patients: those with impaired mobility of laryngeal structures on ultrasound, those without impaired mobility.
To visualise arytenoid motion in subjects with shadow artifact using the standard dTLUS approach, by optimising dTLUS acquisitions including curvilinear probe acquisitions, gel cushion acquisitions and lateral mode acquisitions. | 6 months
  - Sensitivity and specificity for the prediction of a recovery for each quantitative index proposed before the start of speech therapy on the population tested."

CONTACTS AND LOCATIONS:
Overall Officials: Christophe TRESALLET, Pr, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris